CLINICAL TRIAL: NCT03434808
Title: Generation of an Induced Pluripotent Stem (iPS) Cell Bank Immune Matched to a Majority of the US Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: Cellular Dynamics International, Inc. - A FUJIFILM Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-CDI
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: iPS Cell Manufacture and Banking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Whole Blood Donation — Study subjects will provide 250ml whole blood donation for the manufacture and banking of iPS cells.

SUMMARY:
The purpose of this study is to develop a collection of iPS cells called a bank ("Bank") that are immune-matched to a large percentage of the US population by containing the most common HLA haplotypes in the US population.

DETAILED DESCRIPTION:
This study is being done to produce a bank of iPS cells that researchers from around the world can use for many different purposes. Some examples of such uses include basic research, discovery of new medicines, developing new products and services useful for studying human disease, and developing new cell-based products useful for treating people that have diseases. The idea of using cells made from human iPS cells to treat human diseases is of great interest in medicine. In this bank, a single donor's cells could be used to treat many people.

The iPS cells that are made as part of this study will be included in a bank owned by CDI. The iPS cells and the cells made from them will be available for laboratory research or for clinical use in patients. It is possible that the iPS cells made from the blood donated and cells made from the iPS cells could be beneficial to many different patients and be used for many different research projects to understand human biology and disease.

ELIGIBILITY:
Inclusion Criteria:

1. Be associated with an NMDP/Be The Match-operated donor center or non-operated donor center that has an IRB Authorization Agreement with the NMDP IRB and allows NMDP staff to directly contact their donors
2. Possess an HLA haplotype of interest to the Study
3. Be at least 18 years of age and not past 61st birthday
4. Meet the following criteria and requirements:

4.1 Meet the donor requirements under 21 CFR 1271 and related August 2007 guidance 4.2 Body weight of at least 110 pounds 4.3 Complete and pass the abbreviated Health History Screening questionnaire 4.4 Complete and pass the full Health History questionnaire after donor enrollment 4.5 Non-reactive for any FDA-listed relevant communicable disease agent 4.6 Non-reactive for cytomegalovirus (CMV) 4.7 Express blood group O

Exclusion Criteria:

1. Be unwilling or unable to give informed consent
2. Be pregnant
3. Have a prior history of: (i) a bone marrow transplant, or (ii) cancer of any type

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Twelve whole blood samples donated for the manufacture and banking of iPS cells | 2 years
  The objective will have been met when donor blood samples have been collected from eligible donors possessing homozygous HLA haplotypes of interest providing a beneficial match to at least 95 percent of the US population as determined by the matching algorithm used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Confer, MD, Principal Investigator — National Marrow Donor Program; Amanda Mack, PhD, Principal Investigator — Cellular Dynamics International, Inc. - A FUJIFILM Company

IPD SHARING:
Plan to Share IPD: No